CLINICAL TRIAL: NCT04249206
Title: Outcome of Endodontic Treatment in Patient Treated With a Hydraulic Sealer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cittadella Universitaria (Other)
Responsible Party: Principal Investigator, Giulia Bardini, Principal Investigator, Cittadella Universitaria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETEBCB
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Apical Periodontitis
Keywords: root canal obturation; hydraulic sealer; single cone; endodontic outcome
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydraulic Sealer Group (Experimental): The single-cone obturation technique is based on a master cone of gutta-percha in conjunction with a hydraulic sealer.
  Hydraulic endodontic cements exhibit excellent hydraulic properties, biocompatibility and bioactivity.
  Interventions: Procedure: Root Canal Treatment
- Zinc oxide-eugenol Sealer Group (Active Comparator): The continuous wave of condensation of gutta-percha and a zinc oxide-eugenol (ZOE) sealer is a gold standard in endodontic obturation.
  Interventions: Procedure: Root Canal Treatment

INTERVENTIONS:
Procedure: Root Canal Treatment

SUMMARY:
The objective of the study is to evaluate and compare, clinically and radiographically, the outcome of non surgical primary/secondary root canal treatment using a hydraulic sealer or a zinc oxide-eugenol sealer.

ELIGIBILITY:
Inclusion Criteria:

* a permanent, single or multi-rooted mature tooth
* clinical diagnosis of irreversible pulpitis
* diagnosis of apical periodontitis

Exclusion Criteria:

* subjects with immune-compromised status
* subjects with an overall poor prognosis for their treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Periapical Healing | 4 year
  Clinical and radiographic evidence of the absence of apical periodontitis or healing of each tooth (PAI score <2)

SECONDARY OUTCOMES:
tooth survival | 4 year
  Success was defined if the tooth was asymptomatic and considered to be functional regardless of its PAI score

REFERENCES:
- [Derived] Bardini G, Casula L, Ambu E, Musu D, Mercade M, Cotti E. A 12-month follow-up of primary and secondary root canal treatment in teeth obturated with a hydraulic sealer. Clin Oral Investig. 2021 May;25(5):2757-2764. doi: 10.1007/s00784-020-03590-0. Epub 2020 Sep 28. PMID 32989597